CLINICAL TRIAL: NCT02142543
Title: The Effect of 2-DeNT Oral Topical Powder on Minor Recurrent Aphthous Ulcer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BCDOrtho1; 2011-23-BCD (Other: IRB number)
Record Dates: First submitted 2014-04-24; First posted 2014-05-20 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Minor Recurrent Aphthous Stomatitis Lesions
MeSH Terms: interventions — Karaya Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo powder containing zinc oxide, karaya gum, and yellow dye, which was added to imitate the color of the original powder, applied twice a day until the ulcer had resolved, an expected average of 3-5 days
  Interventions: Drug: Placebo Comparator
- 2-DeNT powder (Experimental): 2-DeNT powder containing dexamethasone, diphenhydramine, tetracycline, metronidazole, nystatin, zinc oxide, and karaya gum, applied twice a day until the ulcer had resolved, applied twice a day until the ulcer had resolved, in an expected average of 3 to 5 days
  Interventions: Drug: 2-DeNT powder

INTERVENTIONS:
Drug: 2-DeNT powder — powder included dexamethasone, diphenhydramine, tetracycline, metronidazole, nystatin, zinc oxide, and karaya gum
  Arms: 2-DeNT powder
Drug: Placebo Comparator
  Other Names: placebo powder containing zinc oxide, karaya gum, and yellow dye, which was added to imitate the color of the original powder
  Arms: placebo

SUMMARY:
This is a prospective, randomized, blinded, placebo-controlled, crossover clinical trial to evaluate the efficacy of 2-DeNT oral topical powder in the treatment of recurrent aphthous stomatitis (RAS). To be included in the study, subjects must have had minor RAS ulcers of less than 48 hours duration. It was randomly determined which powder was used first; all subjects used both the 2-DeNT powder and the placebo powder. Subjects applied the powder twice daily and maintained a daily log recording the size of the ulcer, its erythema score, and their level of pain. The subjects continued applying the 2-DeNT powder until the ulcer was resolved.

ELIGIBILITY:
Inclusion Criteria:

* a history of minor recurrent aphthous stomatitis (RAS) lesions occurring at least 3-4 time/ year, and usually requiring 5 or more days to resolve
* presence of an active ulcer of less than 48 hours duration on either the buccal or labial mucosa (making them more easily accessible for powder application)
* willing and able to give informed consent

Exclusion Criteria:

* pregnant or lactating
* if ulcers were manifestations of a systemic disease process such as ulcerative colitis, Crohn's disease, Behcet's syndrome, or anemia;
* concurrent clinical conditions that could either pose a health risk to the patient by being involved in the study or potentially influence the outcome of the study
* hypersensitivity to dexamethasone, diphenhydramine, tetracycline, metronidazole, nystatin, karaya gum, or zinc oxide
* having used corticosteroids, oral retinoids, or other immunomodulatory agents within one month of participation in the study; non-steroidal anti-inflammatory agents (e.g., aspirin, ibuprofen, etc.), acetaminophen, or oral antihistamines chronically within one month of participation in the study or any use within five days of participation in the study; topical medication (including steroids, retinoids, and anti-microbial drugs) within two weeks of participation in the study, systemic antibiotics within two weeks of participation in the study; any preparation or medication (OTC or prescription) applied to the ulcer within 48 hours of participation in the study
* history of drug or alcohol abuse
* having had any dental work within 2 weeks of study entry
* having had any orthodontic or oral appliances (that could cause oral trauma) within 1 cm of the ulcer or any recollection of trauma in the area of the ulcer
* participating in any other study involving investigational or marketed products within 1 month of study entry or plans to participate in such an investigation during this study.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Ulcer size | From time of randomization until ulcer was healed, an expected average of 3 to 5 days
  Size was measured from the outside edge of the white border to the outside edge of the opposite white border. If the ulcer was oval in shape, its longest dimension was measured.

SECONDARY OUTCOMES:
Erythema | From time of randomization until ulcer was healed, an expected average of 3 to 5 days
  Erythema levels were recorded on a scale of 0 to 4 (0= no redness, 1= faint redness, 2= light red/pink, 3= moderate redness, 4= severe redness) using a guide that provided both picture and word descriptions of the degree of redness associated with each number on the scale

OTHER OUTCOMES:
Pain | From time of randomization until ulcer was healed, an expected average of 3 to 5 days
  The perceived level of pain or discomfort was noted by the subject using a 10 cm visual analogue scale (VAS) with anchors of "no pain" and "worst pain ever"

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M Baylor College of Dentisry, Dallas, Texas, United States